CLINICAL TRIAL: NCT02776644
Title: CLINICAL OUTCOME OF ADVANCED RENAL CELL CARCINOMA IN TAIWAN, A RETROSPECTIVE NHIA DATABASE ANALYSIS
Brief Title: Clinical Outcome Of Advanced Renal Cell Carcinoma In Taiwan
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: A6181222
Record Dates: First submitted 2016-05-11; First posted 2016-05-18 (Estimated); Results first posted 2019-04-29 (Actual); Last update posted 2023-03-16 (Actual); Status verified 2019-04

CONDITIONS: Renal Cell Carcinoma
Keywords: renal cell carcinoma; sunitinib, pazopanib; temsirolimus; sorafenib; everolimus; interferon alpha; interleukin 2
MeSH Terms: conditions — Carcinoma, Renal Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The clinical outcome of advanced / metastatic renal cell carcinoma has been changed since targeted therapy being widely applied. This study will retrospectively analyse the clinical outcome of advanced renal cell carcinoma captured in Taiwan National Health Insurance Research Database.

DETAILED DESCRIPTION:
Targeted therapy agents have significantly changed the clinical outcome of advanced / metastatic renal cell carcinoma. However, the dosing pattern varied and might result in impact to duration of treatment. In Taiwan, National Health Insurance system has a coverage more than 90% of population and thus can serve as an appropriate database for further analysis on Taiwanese advanced renal cell carcinoma. This study will retrospectively analyse the clinical outcome of advanced renal cell carcinoma captured in Taiwan National Health Insurance Research Database.

ELIGIBILITY:
Inclusion Criteria:

* advanced/metastatic renal cell carcinoma

Exclusion Criteria:

* N/A

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: advanced/metastatic renal cell carcnioma
Sampling Method: Non-Probability Sample
Enrollment: 1349 (Actual)
Dates: Start 2016-10-15 (Actual); Primary Completion 2017-12-30 (Actual); Study Completion 2017-12-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A6181222&StudyName=Clinical+Outcome+Of+Advanced+Renal+Cell+Carcinoma+In+Taiwan%2C+A+Retrospective+Nhia+Database+Analysis

RESULTS

PARTICIPANT FLOW:
Groups:
- Sunitinib: Participants who were diagnosed with metastatic renal cell carcinoma (RCC), as per the records of Catastrophic illness patient database and National health insurance research database (NHIRD) (from January 2004 to December 2015), and were treated with Sunitinib capsule 12.5 milligram (mg), were included in this study and their data was observed retrospectively.
- Pazopanib: Participants who were diagnosed with metastatic RCC, as per the records of Catastrophic illness patient database and NHIRD (from January 2004 to December 2014), and were treated with Pazopanib tablets 200 mg, were included in this study and their data was observed retrospectively.
Period: Overall Study
Arm/Group | Sunitinib | Pazopanib
Started | 1223 | 126
Completed | 1223 | 126
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: All Taiwanese participants diagnosed with metastatic RCC during the time period of January 2004 to December 2015 and received treatment (Sunitinib or Pazopanib).
Groups:
- Total: Total of all reporting groups
Arm/Group | Sunitinib | Pazopanib | Total
Number analyzed (Participants) | 1223 | 126 | 1349
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.14 (13) | 66.45 (12.95) | 64.33 (12.99)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 318 | 37 | 355
  Male | 903 | 89 | 992
  Unknown | 2 | 0 | 2
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Participants by Different Income Levels [Count of Participants; unit: Participants] — Income levels of the participants were divided into three categories, 1) Low income, which included all the participants with income less the 15,000 new Taiwan dollars per month, 2) Median income, which included all the participants with income 15,000-24,999 new Taiwan dollars per month, 3) High income, which included all the participants with income more than 25,000 new Taiwan dollars per month.
  Participants
    Low income | 279 | 24 | 303
    Medium income | 351 | 37 | 388
    High income | 593 | 65 | 658
Participants With Different Co-Morbid Conditions [Count of Participants; unit: Participants] — Co-morbid conditions included all diseases (hypertension, diabetes mellitus, dyslipidemia, coronary artery disease, chronic kidney disease, and liver cirrhosis) other than metastatic RCC, from which the participants were suffering during the observation period. A participant could have more than one co-morbid condition. Here, NHIRD in the comment field signifies to National Health Insurance Research Database.
  Participants
    Hypertension | 634 | 59 | 693
    Diabetes mellitus | 350 | 39 | 389
    Dyslipidemia | 312 | 32 | 344
    Coronary artery disease | 188 | 30 | 218
    Chronic kidney disease | 159 | 17 | 176
    Liver cirrhosis | 26 | NA — Due to NHIRD regulation, data cannot be reported if sample size less than equal to (<=) 3. | NA — Total not calculated because data are not available (NA) in one or more arms.
Participants Who Had Received Concomitant-Medications [Count of Participants; unit: Participants] — Concomitant-medications were the medications that the study participants had taken along with Sunitinib or Pazopanib. Participants could have received more than one concomitant medication.
  Participants
    Beta blockers | 364 | 38 | 402
    Calcium channel blockers | 543 | 57 | 600
    Diuretics | 331 | 38 | 369
    Angiotensin-converting enzyme inhibitors | 135 | 11 | 146
    Angiotensin receptor blocker | 397 | 40 | 437
    Insulin | 53 | 7 | 60
    Biguanides | 189 | 22 | 211
    Sulfonylurea | 186 | 16 | 202
    Glucosidase inhibitors | 56 | 4 | 60
    Thiazolidinediones | 46 | NA — Due to NHIRD regulation, data cannot be reported, if sample size <=3. | NA — Total not calculated because data are not available (NA) in one or more arms.
    Dipeptidyl peptidase 4 inhibitors | 80 | 19 | 99
    Statins | 242 | 27 | 269
    Fibrates | 56 | 6 | 62
    Bile acid sequestrants and Nicotinic acid | 4 | NA — Due to NHIRD regulation, data cannot be reported, if sample size <=3. | NA — Total not calculated because data are not available (NA) in one or more arms.
    Ezetimibe | 18 | NA — Due to NHIRD regulation, data cannot be reported, if sample size <=3. | NA — Total not calculated because data are not available (NA) in one or more arms.
    Antiplatelets | 352 | 34 | 386
    Anticoagulants | 32 | NA — Due to NHIRD regulation, data cannot be reported, if sample size <=3. | NA — Total not calculated because data are not available (NA) in one or more arms.
Participants Admitted/Visited to Hospital by Type of Hospitals [Count of Participants; unit: Participants] — Medical center was defined by Taiwan Food and Drug Administration as hospitals accredited with medical training, research, high-tech equipment, and ability to support other hospital nearby.
  Participants
    Medical center | 865 | 91 | 956
    Other than medical center | 358 | 35 | 393
Participants Admitted/Visited to the Hospital According to the Geographical Location of Hospitals [Count of Participants; unit: Participants] — Geographical location of hospitals included capital area and non-capital area. Capital area hospitals includes the hospitals that were located at national capital and non-capital area hospitals includes the hospitals that were located outside of national capital.
  Participants
    Capital area hospital | 447 | 40 | 487
    Non-capital area hospital | 776 | 86 | 862

OUTCOME MEASURES:

1. Primary Outcome: Duration of Sunitinib and Pazopanib Treatment in Participants
Description: Treatment durations (in days) of Sunitinib and Pazopanib were calculated from the date of the first prescription to the last dose of Sunitinib and Pazopanib during the 11 year observation period.
Time Frame: during the observation period of 11 years
Population: as for baseline characteristics
Measure: Median (Full Range); unit: days
Arm/Group | Sunitinib | Pazopanib
Number analyzed (Participants) | 1223 | 126
days | 171 [1 to 2153] | 114.5 [1 to 1219]

2. Primary Outcome: Cumulative Number of Capsules of Sunitinib and Pazopanib Administered From the Time of Start of Treatment Up to Month 3
Description: The cumulative number of Sunitinib and Pazopanib capsules which were given to the participants from the time of start of treatment up to Month 3 were reported here.
Time Frame: from the time of start of treatment up to Month 3
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: capsules
Arm/Group | Sunitinib | Pazopanib
Number analyzed (Participants) | 1223 | 126
capsules | 190.1 (81.5) | 215.1 (118.4)

3. Primary Outcome: Cumulative Number of Capsules of Sunitinib and Pazopanib Administered From Month 3 to Month 6
Description: The cumulative number of Sunitinib and Pazopanib capsules which were given to the participants from Month 3 (after the start of treatment) to Month 6 were reported here.
Time Frame: Month 3 up to Month 6
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: capsules
Arm/Group | Sunitinib | Pazopanib
Number analyzed (Participants) | 1223 | 126
capsules | 165.0 (88.4) | 193.2 (118.9)

4. Primary Outcome: Cumulative Number of Capsules of Sunitinib and Pazopanib Administered From Month 6 to Month 9
Description: The cumulative number of Sunitinib and Pazopanib capsules which were given to the participants from Month 6 (after the start of treatment) to Month 9 were reported here.
Time Frame: Month 6 up to Month 9
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: capsules
Arm/Group | Sunitinib | Pazopanib
Number analyzed (Participants) | 1223 | 126
capsules | 174.9 (83.5) | 186.5 (111.1)

5. Primary Outcome: Cumulative Number of Capsules of Sunitinib and Pazopanib Administered From Month 9 to Month 12
Description: The cumulative number of Sunitinib and Pazopanib capsules which were given to the participants from Month 9 (after the start of treatment) to Month 12 were reported here.
Time Frame: Month 9 up to Month 12
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: capsules
Arm/Group | Sunitinib | Pazopanib
Number analyzed (Participants) | 1223 | 126
capsules | 176.5 (83.4) | 212.1 (109.9)

6. Primary Outcome: Cumulative Number of Capsules of Sunitinib and Pazopanib Administered From the Time of Start of Treatment Up to Month 12
Description: The cumulative number of Sunitinib and Pazopanib capsules which were given to the participants from the time of start of treatment to Month 12 were reported here.
Time Frame: from the time of start of treatment up to Month 12
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: capsules
Arm/Group | Sunitinib | Pazopanib
Number analyzed (Participants) | 1223 | 126
capsules | 435.4 (326.8) | 438.0 (375.1)

7. Primary Outcome: Overall Renal Cell Carcinoma (RCC) Related Direct Medical Cost From the Diagnosis Date to the First Dose of Sunitinib and Pazopanib
Description: Direct medical costs include the cost of the Sunitinib or Pazopanib and all follow-up costs for other medication and health care interventions in ambulatory, inpatient, and nursing care. All specialist and general practitioner care, including emergency care, as well as rehabilitation and physiotherapy.
Time Frame: from the time of disease diagnosis till the first dose of Sunitinib and Pazopanib
Population: All Taiwanese participants diagnosed with metastatic RCC during the time period of January 2004 to December 2015 and received treatment (Sunitinib or Pazopanib). Overall number of participants analyzed signifies participants who were evaluable for this outcome measure.
Measure: Number; unit: new Taiwan dollars
Arm/Group | Sunitinib | Pazopanib
Number analyzed (Participants) | 1221 | 126
new Taiwan dollars | 176,969,380 | 45,442,288

8. Primary Outcome: Overall Renal Cell Carcinoma (RCC) Related Direct Medical Cost From the First Dose of the Sunitinib and Pazopanib to the End of Observation Period
Description: as for outcome 7
Time Frame: From first dose of drug to the end of observation period (up to 11 years)
Population: as for outcome 7
Measure: Number; unit: new Taiwan dollars
Arm/Group | Sunitinib | Pazopanib
Number analyzed (Participants) | 1221 | 126
new Taiwan dollars | 1,519,649,383 | 78,745,896

9. Primary Outcome: Overall Survival
Description: Overall survival of participants was defined as time (in days) between date of prescribing treatment (Sunitinib or Pazopanib) till date of death.
Time Frame: from the time of first prescription of Sunitinib or Pazopanib till date of death (during the observation period of 11 years)
Population: as for baseline characteristics
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Sunitinib | Pazopanib
Number analyzed (Participants) | 1223 | 126
days | 490 [443 to 536] | 416 [312 to 807]

10. Primary Outcome: Number of Participants With Changes in Prescription Patterns of Antihypertensive Medication From the Time of First Dose of Drug at Month 1
Description: Changes in the prescription patterns of antihypertensive medication were categorized as: 1) Unchanged: no change in the count/number of capsules or class(es) of the antihypertensive medication at Month 1 as compared to the time of first dose, 2) Increased: increase in counts/number of capsules of the ongoing class(es) of the antihypertensive medication at Month 1 as compared to the time of first dose, 3) Decreased: Decrease in the counts/number of capsules of ongoing class(es) of antihypertensive medication at Month 1 as compared to the time of first dose, 4) Switched: shifted to other class(es) of antihypertensive medication without changes in counts of antihypertensive medication at Month 1 as compared to the time of first dose. The number of participants with change in prescription patterns based on the specified categories is reported.
Time Frame: time of first dose of the drug, Month 1
Population: All Taiwanese participants diagnosed with metastatic RCC during the time period of January 2004 to December 2015 and received treatment (Sunitinib or Pazopanib). Here, Overall number of participants analyzed signifies participants who were evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Sunitinib | Pazopanib
Number analyzed (Participants) | 189 | 43
Participants
  Unchanged | 96 | 9
  Increased | 85 | 14
  Decreased | 63 | 14
  Switched | 35 | 6

11. Primary Outcome: Number of Participants With Changes in Prescription Patterns of Antihypertensive Medication From the Time of First Dose of Drug at Month 3
Description: Changes in the prescription patterns of antihypertensive medication were categorized as: 1) Unchanged: no change in the count/number of capsules or class(es) of the antihypertensive medication at Month 3 as compared to the time of first dose, 2) Increased: increase in counts/number of capsules of the ongoing class(es) of the antihypertensive medication at Month 3 as compared to the time of first dose, 3) Decreased: Decrease in the counts/number of capsules of ongoing class(es) of antihypertensive medication at Month 3 as compared to the time of first dose, 4) Switched: shifted to other class(es) of antihypertensive medication without changes in counts of antihypertensive medication at Month 3 as compared to the time of first dose. The number of participants with change in prescription patterns based on the specified categories is reported.
Time Frame: time of first dose of the drug, Month 3
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | Sunitinib | Pazopanib
Number analyzed (Participants) | 421 | 61
Participants
  Unchanged | 142 | 20
  Increased | 176 | 21
  Decreased | 57 | 13
  Switched | 46 | 7

12. Primary Outcome: Number of Participants With Changes in Prescription Patterns of Antihypertensive Medication From the Time of First Dose of Drug at Month 6
Description: Changes in the prescription patterns of antihypertensive medication were categorized as: 1) Unchanged: no change in the count/number of capsules or class(es) of the antihypertensive medication at Month 6 as compared to the time of first dose, 2) Increased: increase in counts/number of capsules of the ongoing class(es) of the antihypertensive medication at Month 6 as compared to the time of first dose, 3) Decreased: Decrease in the counts/number of capsules of ongoing class(es) of antihypertensive medication at Month 6 as compared to the time of first dose, 4) Switched: shifted to other class(es) of antihypertensive medication without changes in counts of antihypertensive medication at Month 6 as compared to the time of first dose. The number of participants with change in prescription patterns based on the specified categories is reported.
Time Frame: the first dose of the drug, Month 6
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | Sunitinib | Pazopanib
Number analyzed (Participants) | 442 | 64
Participants
  Unchanged | 132 | 18
  Increased | 213 | 24
  Decreased | 54 | 11
  Switched | 43 | 11

13. Primary Outcome: Number of Participants With Changes in Prescription Patterns of Antihypertensive Medication From the Time of First Dose of Drug at Month 12
Description: Changes in the prescription patterns of antihypertensive medication were categorized as: 1) Unchanged: no change in the count/number of capsules or class(es) of the antihypertensive medication at Month 12 as compared to the time of first dose, 2) Increased: increase in counts/number of capsules of the ongoing class(es) of the antihypertensive medication at Month 12 as compared to the time of first dose, 3) Decreased: Decrease in the counts/number of capsules of ongoing class(es) of antihypertensive medication at Month 12 as compared to the time of first dose, 4) Switched: shifted to other class(es) of antihypertensive medication without changes in counts of antihypertensive medication at Month 12 as compared to the time of first dose. The number of participants with change in prescription patterns based on the specified categories is reported.
Time Frame: the first dose of the medication, Month 12
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | Sunitinib | Pazopanib
Number analyzed (Participants) | 446 | 66
Participants
  Unchanged | 104 | 17
  Increased | 262 | 28
  Decreased | 47 | 10
  Switched | 33 | 11

14. Primary Outcome: Number of Participants Who Received Antihypertensive Medication at Baseline
Description: To calculate number of patient receiving antihypertensive prescriptions at baseline for each TKI users and classify the patterns of changes into unchanged, switched, increased and decreased. Shifting to other class(es) of antihypertensive agents without changes in counts of antihypertensive medication is defined as being switched.
Time Frame: Baseline (at the beginning of 11 year observation period)
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | Sunitinib | Pazopanib
Number analyzed (Participants) | 657 | 94
Participants | 518 | 77

15. Primary Outcome: Number of Participants Who Received Antihypertensive Medication From Baseline to Month 1
Description: To calculate number of patient receiving antihypertensive prescriptions at Month 1 for each TKI users and classify the patterns of changes into unchanged, switched, increased and decreased. Shifting to other class(es) of antihypertensive agents without changes in counts of antihypertensive medication is defined as being switched.
Time Frame: Baseline (at the beginning of 11 year observation period) up to Month 1
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | Sunitinib | Pazopanib
Number analyzed (Participants) | 657 | 94
Participants | 66 | 5

16. Primary Outcome: Number of Participants Who Received Antihypertensive Medication From Month 1 to Month 3
Description: To calculate number of patient receiving antihypertensive prescriptions from Month 1 to Month 3 for each TKI users and classify the patterns of changes into unchanged, switched, increased and decreased. Shifting to other class(es) of antihypertensive agents without changes in counts of antihypertensive medication is defined as being switched.
Time Frame: Month 1 up to Month 3 since Sunitinib or Pazopanib initiation (during the observation period of 11 years)
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | Sunitinib | Pazopanib
Number analyzed (Participants) | 657 | 94
Participants | 30 | 7

17. Primary Outcome: Number of Participants Who Received Antihypertensive Medication From Month 3 to Month 6
Description: To calculate number of patient receiving antihypertensive prescriptions from Month 3 to Month 6 for each TKI users and classify the patterns of changes into unchanged, switched, increased and decreased. Shifting to other class(es) of antihypertensive agents without changes in counts of antihypertensive medication is defined as being switched.
Time Frame: Month 3 up to Month 6 since Sunitinib or Pazopanib initiation (during the observation period of 11 years)
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | Sunitinib | Pazopanib
Number analyzed (Participants) | 657 | 94
Participants | 15 | 5

18. Primary Outcome: Number of Participants Who Received Antihypertensive Medication From Month 6 to Month 12
Description: To calculate number of patient receiving antihypertensive prescriptions from Month 6 to Month 12 for each TKI users and classify the patterns of changes into unchanged, switched, increased and decreased. Shifting to other class(es) of antihypertensive agents without changes in counts of antihypertensive medication is defined as being switched.
Time Frame: Month 6 up to Month 12 since Sunitinib or Pazopanib initiation (during the observation period of 11 years)
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | Sunitinib | Pazopanib
Number analyzed (Participants) | 657 | 94
Participants | 18 | NA — Due to NHIRD regulation, data cannot be reported if sample size <=3.

ADVERSE EVENTS:
Description: Due to the non-interventional nature of this study, adverse events (AEs) were not collected for this study.
Arm/Group | Sunitinib | Pazopanib
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
Prioritization of outcome measures as primary and secondary was based on the study team's discretion.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-08-31): https://cdn.clinicaltrials.gov/large-docs/44/NCT02776644/Prot_SAP_000.pdf